CLINICAL TRIAL: NCT02598284
Title: Midwest Small Practice Care Transformation Research Alliance (MSPCTRA)
Brief Title: Healthy Hearts in the Heartland
Acronym: H3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Alliance of Chicago Community Health Services (Other); American Medical Association (Other); Illinois Department of Public Health (Other); MetaStar, Inc. (Industry); Northern Illinois University (Other); Northwestern Medical Group (Other); Purdue University (Other); Telligen, Inc. (Industry); University of Chicago (Other)
Responsible Party: Principal Investigator, Abel Kho, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HS 023921-01
Record Dates: First submitted 2015-10-15; First posted 2015-11-05 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Cardiovascular Diseases
Keywords: Preventive measures; Quality Improvement
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Point-of-Care Systems; Population Health Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Point of Care (POC) Only (Experimental): Clinics will receive facilitation to implement point-of-care (POC) quality improvement strategies to accelerate performance on ABCS clinical measures. All strategies will focus on aspects of the clinical encounter.
  Interventions: Other: Point of Care
- POC + Population Managment (PM) (Experimental): Clinics will receive facilitation to implement point-of-care (POC) quality improvement strategies as well as population management (PM) strategies to accelerate performance on ABCS clinical measures. Strategies in this arm will occur both at the clinical encounter and strategies aimed at the time between clinical encounters.
  Interventions: Other: Point of Care; Other: Population Management

INTERVENTIONS:
Other: Point of Care — Practice facilitators will work with practices to implement strategies to improve ABCS care during the patient encounter. Some examples of these types of quality improvement initiatives are electronic reminders and clinical decision support to prescribe aspirin or a statin at the time of a visit, improving how your practice collects blood pressure measures to increase clinicians' willingness to act on readings, or electronic reminders for nursing staff that there is no lipid panel in record and have a standing order to act on this.
Other: Population Management — Practice Facilitators will work with practices to both implement Point of Care strategies as well as population management strategies. These practices will use their EHR and/or receive training to use the popHealth software package, which works with data from the EHR, to generate lists of high-risk patients that need outreach for one of the ABCS domains (such as conducting outreach to patients who are not on aspirin who would benefit from this therapy).
  Practices in this arm will receive the opportunity to link to community resources such as pharmacists who could assist patients with medication management or tobacco quit lines through the HealtheRx program.
  Arms: POC + Population Managment (PM)

SUMMARY:
This study evaluates the ability of small primary care practices to 1) implement point-of-care and population management quality improvement strategies to improve cardiovascular quality of care (e.g., clinical decision support, patient education and counseling, or referral to smoking quit lines), and 2) implement the PopHealth performance measurement software to evaluate performance on the ABCS (aspirin when appropriate, blood pressure control, cholesterol management, and when applicable, smoking cessation) and allow regional benchmarking. This minimal risk study is a practice-randomized trial to determine a) whether point of care strategies improve ABCS performance measures compared to baseline, and b) whether adding locally tailored population management strategies to POC strategies improves performance on the ABCS measures more than POC strategies alone.

DETAILED DESCRIPTION:
The investigators specific aims are to:

1. Evaluate the ability of small practices in the investigators region to 1) implement point-of-care (POC) and population management (PM) quality improvement strategies to improve the ABCS, and 2) implement the popHealth quality measurement software to evaluate performance on the ABCS and allow regional benchmarking.
2. Conduct a practice-randomized trial to determine a) whether POC strategies improve ABCS performance measures (i.e. aspirin prescribing, blood pressure control, cholesterol management, and smoking cessation counseling) compared to baseline, and b) whether adding locally-tailored PM strategies to POC strategies improves performance on the ABCS measures more than POC strategies alone.
3. Deploy an open source quality measurement platform (popHealth) to establish a regional QI benchmark based on participating practice ABCS measures and enable longitudinal tracking of electronic clinical quality measures (eCQMs) across the investigators region. The investigators will perform a mixed-methods evaluation to examine changes in practices' perceived capacity for quality improvement and whether access to comparative quality data within a region improves the capacity of practices to sustain their quality improvement program around the ABCS and provides a long-term framework for practices to implement new QI activities.

ELIGIBILITY:
Inclusion Criteria:

* Providers practicing in Wisconsin, Illinois, and Indiana.
* Practice is adult primary care-focused; [Further defined: health care organization dedicated to the provision of primary care, and a significant proportion of their patients are adults. Includes, but not limited to, family medicine, general internal medicine, general practice, geriatricians, nurse practitioners and physician assistants.]
* Practice has 20 or fewer primary care providers; [Community health centers with 20 or fewer lead clinicians may be included; multi-specialty practices that provide primary care and have ≤ 20 lead clinicians may be included.]
* Providers must provide informed consent.

Exclusion Criteria:

* Non-English speaking providers

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in appropriate aspirin prescribing from baseline to 12 months | 12 months
  Measured using electronic health record data. Patients age ≥ 18 with eligible encounters during measurement period (year prior and including measurement date) with IVD diagnosis on active problem list (on measurement date) or visit diagnosis (on or within 1 year prior to measurement date) who have aspirin prescribed.
Change in clinical performance on blood pressure control from baseline to 12 months | 12 months
  Measured using electronic health record data. The proportion of adult (age 18-85) patients with hypertension with blood pressure <140/90
Change in clinical performance on cholesterol management from baseline to 12 months | 12 months
  Measured using electronic health record data. The proportion of adult patients who are eligible for statins with a stain prescription on active medication list. Eligible patients for this measure are (1) Patients age ≥ 21 with an ASCVD diagnosis on problem list and (2) Patients age 40-75 with eligible encounters during the study period and diabetes on active problem list or as a visit diagnosis.
Change in clinical performance on smoking cessation from baseline to 12 months | 12 months
  Measured using electronic health record data. The proportion of patients ≥ 18 with eligible encounters during the study period who have an assessment of tobacco use recorded. Then, among patients who report using tobacco, the proportion who have received a tobacco cessation intervention.

SECONDARY OUTCOMES:
Capacity for Quality Improvement | 12 months
  Collected via Change Process Capability Questionnaire (CPCQ)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - Northern Illinois University (NIU), DeKalb, Illinois
  - Telligen, Oak Brook, Illinois
  - Purdue University, West Lafayette, Indiana
  - MetaStar, Madison, Wisconsin

REFERENCES:
- [Derived] Ross SM, Wang A, Anthony L, Persell SD, Yu J, Kho AN. Is more better? The impact of implementing more interventions for hypertension control in a practice facilitation study for small- and medium-sized practices. J Hum Hypertens. 2023 Nov;37(11):1007-1014. doi: 10.1038/s41371-023-00813-1. Epub 2023 Mar 22. PMID 36949284
- [Derived] Ciolino JD, Jackson KL, Liss DT, Brown T, Walunas TL, Murakami L, Chung I, Persell SD, Kho AN. Design of healthy hearts in the heartland (H3): A practice-randomized, comparative effectiveness study. Contemp Clin Trials. 2018 Aug;71:47-54. doi: 10.1016/j.cct.2018.06.004. Epub 2018 Jun 2. PMID 29870868